CLINICAL TRIAL: NCT01369316
Title: Circumferential Submucosal Incision Endoscopic Mucosal Resection Versus Conventional Endoscopic Resection for the Removal of Large Laterally Spreading Tumours and Sessile Polyps of the Colon
Brief Title: Circumferential Submucosal Incision Endoscopic Mucosal Resection Versus Conventional Endoscopic Mucosal Resection of Colonic Polyps
Acronym: CSIEMR
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: study abandoned
Sponsor: Professor Michael Bourke (Other)
Responsible Party: Sponsor-Investigator, Professor Michael Bourke, Dr Michael Bourke, Western Sydney Local Health District
Organization: Western Sydney Local Health District (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EMR-002-CSI
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Colonic Polyps
MeSH Terms: conditions — Colonic Polyps | interventions — Endoscopic Mucosal Resection

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Circumferential Submucosal Incision Resection (Experimental)
  Interventions: Procedure: Circumferential Submucosal Incision Resection
- Endoscopic Mucosal Resection (Active Comparator): Patients randomised into this arm will receive the conventional treatment Endoscopic Mucosal Resection in which the sessile lesion is injected and snared by piecemeal technique.
  Interventions: Procedure: Endoscopic Mucosal Resection

INTERVENTIONS:
Procedure: Circumferential Submucosal Incision Resection — The patient is randomized, if in the active arm the procedure will continue as Circumferential Submucosal Incision Endoscopic Mucosal Resection.
  Arms: Circumferential Submucosal Incision Resection
Procedure: Endoscopic Mucosal Resection — Patients randomised into this Intervention type will have Endoscopic Mucosal Resection performed
  Arms: Endoscopic Mucosal Resection

SUMMARY:
That Circumferential Submucosal Incision Endoscopic Mucosal Resection (CSI-EMR) will be at least as safe but more effective than conventional EMR for injection assisted EMR of large laterally spreading tumour and sessile polyps of the colon.

DETAILED DESCRIPTION:
The investigators have recently developed a new, and the investigators believe safer and more effective technique for endoscopic mucosal resection (EMR). Utilising the new method the investigators make small cuts around the polyp to isolate it. Subsequently the Gelofusine solution is injected beneath the polyp and provides greater elevation. This allows us to improve the chance of removal of the entire polyp with one attempt in one piece. It is preferable to remove the polyp in one piece as it minimises the chance of leaving residual polyp tissue behind. Our team has recently completed an animal study comparing our newly developed technique to conventional EMR. The investigators have found significant improvements in our ability to completely remove the polyp in one attempt. There have also been recent studies overseas that have shown this new technique to be quite effective.

ELIGIBILITY:
Inclusion Criteria:

* Can give informed consent to trial participation
* Age greater than 18
* Adenomas that have not have previously been attempted for resection (i.e. naïve lesions)
* Adenoma size greater than 20 mm

Exclusion Criteria:

* Age less than 18
* Previous resection or attempted resection of target adenoma lesion
* Pregnant patients

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-09 (Actual); Primary Completion 2020-03-09 (Actual); Study Completion 2020-03-09 (Actual)

PRIMARY OUTCOMES:
Efficacy of CSI EMR (Rates of en-bloc resection, recurrence rates) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Michael J Bourke, Principal Investigator — Westmead Hospital - Endoscopy Unit
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia